CLINICAL TRIAL: NCT05847582
Title: Pilot RCT to Evaluate Feasibility and Acceptability of mSTARS
Brief Title: mHealth-supported Skills Training for Alcohol-Related Suicidality Phase 3
Acronym: mSTARS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00113104_1
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Drinking; Suicide
MeSH Terms: conditions — Alcohol Drinking; Suicide | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mSTARS (Experimental): Participants randomized to the mSTARS condition will receive standard inpatient care while hospitalized at Duke. They will also receive an intervention that combines inpatient skills training and the mHealth telephone app. Inpatient emotional regulation skills training will be completed while participants are receiving inpatient treatment at Duke. Upon discharge from Duke, patients will download the mHealth app on their personal phones to use in their personal environments for 30 days. The app is designed to encourage participants to apply skills acquired in inpatient skills training to real-life situations.
  Interventions: Behavioral: Standard inpatient psychiatric care; Behavioral: Inpatient Skills Training; Behavioral: mHealth-supported Skills Training for Alcohol-Related Suicidality (mSTARS)
- Treatment As Usual (Active Comparator): Participants randomized to the treatment-as-usual condition will receive standard inpatient care provided at Duke.
  Interventions: Behavioral: Standard inpatient psychiatric care
- Treatment As Usual + Skills Training (Active Comparator): Participants randomized to this condition will receive standard inpatient care and inpatient emotional regulation skills training.
  Interventions: Behavioral: Standard inpatient psychiatric care; Behavioral: Inpatient Skills Training

INTERVENTIONS:
Behavioral: Standard inpatient psychiatric care — All participants involved in this study will receive standard of care treatment at Duke University Medical Center's Behavioral Health Inpatient Program.
Behavioral: Inpatient Skills Training — Inpatient skills training will be completed while participants are receiving inpatient treatment at BHIP. Skills training includes content designed to improve emotional regulation skills.
  Arms: Treatment As Usual + Skills Training; mSTARS
Behavioral: mHealth-supported Skills Training for Alcohol-Related Suicidality (mSTARS) — mSTARS includes inpatient skills training and a mobile health (mHealth) telephone app designed to encourage participants to apply skills acquired in inpatient skills training to real-life situations.
  Arms: mSTARS

SUMMARY:
Suicide is a high priority public health problem and an increasingly prevalent alcohol-related consequence. One-third of people who die by suicide consume alcohol at hazardous rates in the year preceding death. Most people in an acute suicide crisis who present for treatment are admitted to acute psychiatric hospitalization. Yet, the 30-day period following discharge from hospitalization is by far the riskiest period for another suicide crisis. The specific aim for this project is to evaluate the feasibility and acceptability of an intervention called mHealth-supported Skills Training for Alcohol-Related Suicidality (mSTARS). Thirty-five inpatients with suicidal thoughts or behaviors who misuse alcohol will be randomized to one of three study conditions -- mSTARS, treatment as usual, or treatment as usual with skills training.

DETAILED DESCRIPTION:
Suicide is a high priority public health problem and an increasingly prevalent alcohol-related consequence. One-third of people who die by suicide consume alcohol at hazardous rates in the year preceding death. [Most people in an acute suicide crisis who present for treatment are admitted to acute psychiatric hospitalization. Yet, the 30-day period following discharge from hospitalization is by far the riskiest period for another suicide crisis, (post-discharge rates of suicide are 600 times the global rate). Critically, 50% of suicidal inpatients report alcohol misuse, which further heightens post-discharge risk for suicide.

Acute psychiatric hospitalization focuses on rapid crisis resolution before discharging patients back into their environments with a referral for outpatient care. Outpatient-based cognitive-behavioral skills training in emotion regulation successfully treats concurrent alcohol misuse and suicidal behavior by targeting deficits in emotion regulation associated with both behaviors. Yet, fewer than 50% of psychiatric inpatients follow up with outpatient care once discharged, and those who seek care are often unable to receive it for weeks. Persistently low use of outpatient therapies coupled with alarming post-discharge rates of suicide represents an urgent quality gap. Alternative strategies for inpatient care that extend treatment into the critical post-discharge period are clearly needed to prevent suicide in psychiatric inpatients who misuse alcohol.

The specific aim for this project is to evaluate the feasibility and acceptability of an intervention called mHealth-supported Skills Training for Alcohol-Related Suicidality (mSTARS). Inpatients (N = 35) with suicidal thoughts or behaviors who misuse alcohol will be randomized to one of three study conditions: 1) mSTARS (n = 15), 2) treatment as usual (TAU) plus skills training (n = 10), or 3) TAU alone (n = 10). Primary outcomes include feasibility (e.g., recruitment, retention) and acceptability (e.g., patient satisfaction). Secondary outcomes include suicidal thoughts/behaviors, alcohol use, skills utilization, and rehospitalization.

Participants will complete four study visits, including consent and screening, inpatient treatment, post-treatment assessment, and a 3-month follow-up assessment. After the screening visit, participants will be block-randomized to one of three study conditions listed in item 1.a. above. All participants will receive standard inpatient care. Participants randomized to the mSTARS condition will also receive an intervention that combines inpatient skills training and the mHealth telephone app. Inpatient skills training will be completed while participants are receiving inpatient treatment at BHIP. Skills training includes content designed to improve emotional regulation skills, including motivational enhancement, emotional awareness and acceptance, thinking flexibly, changing emotions, countering cravings, and relapse prevention. Upon discharge from Duke BHIP, patients will download the mHealth app on their personal phones to use in the personal environments for 30 days. The app is designed to encourage participants to apply skills acquired in inpatient skills training to real-life situations. Participants assigned to the TAU plus skills training will receive standard inpatient care plus the inpatient skills training described above. Participants assigned to the TAU condition will receive standard inpatient care only. All participants will be seen for a post-treatment assessment at 30-days and 3-months post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* hospitalized for suicide crisis at Duke BHIP
* an AUDIT-C score indicating hazardous past-month drinking (4 for men; 3 for women) + a 90-day calendar timeline follow-back (TLFB) indicating a minimum of 3 heavy drinking days per week on average (per NIAAA standards)
* owns a smart phone
* fluent in English.

Exclusion Criteria:

* current psychotic or mania symptoms indicated by the MINI Neuropsychiatric Interview 6.0.(MINI)
* receiving ECT at the time of hospitalization, which could inhibit learning
* engaged in weekly outpatient psychotherapy
* discharging to another high level of psychiatric care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are recruited to participate | 30 days
  This is an indication of feasibility of being able to recruit enough participants in a timely manner into the protocol.
Number of participants who complete the post-treatment visit | 30 days
  Retention will be defined as the number of participants who complete the post-treatment visit that occurs 30 days post-discharge.
Number of participants who rate the intervention a 16 or more on the Client Satisfaction Questionnaire. | 30 days
  Acceptability of treatment will be measured by an 8-item measure designed to evaluate client satisfaction. Scores range from 8 to 32, with higher scores indicating higher satisfaction.
Number of participants who score above threshold (34 or more) on the mHealth Satisfaction Questionnaire | 30 days
  Acceptability of treatment will be measured by a 14-item measure designed to measure usability of mobile health apps. Scores range from 14 to 70. Higher scores indicate higher satisfaction.

SECONDARY OUTCOMES:
Average score on the Beck Scale for Suicidal Ideation | 30 days
  Participants will complete the Beck Scale for Suicidal Ideation, a 19-item scale to assess ideation, plans, and/or intent to suicide. Scores range from 0 to 48, with higher scores indicating higher suicide risk.
Average score on the Beck Scale for Suicidal Ideation | 3-month follow-up
  Participants will complete the Beck Scale for Suicidal Ideation, a 19-item scale to assess ideation, plans, and/or intent to suicide. Scores range from 0 to 48, with higher scores indicating higher suicide risk.
Average number of drinking days | 30 days
  Patients will self-report the number of drinking days in the period between their post-treatment visit and the 3-month follow-up visit.
Average number of drinking days | 3-month follow-up
  Patients will self-report the number of drinking days in the period between their post-treatment visit and the 3-month follow-up visit.
Number of participants who report re-hospitalization to an inpatient psychiatry unit. | 30 days
  Treatment inefficacy will be measured by the number of participants who are re-hospitalized in the 30 day period following their enrollment in the study.
Number of participants who report re-hospitalization to an inpatient psychiatry unit. | 3-month follow-up
  Treatment inefficacy will be measured by the number of participants who are re-hospitalized in the 30 day period following their enrollment in the study.
Number of participants who score above 80 on an emotion regulation scale | 30 days
  Number of participants who score above 80 on an emotion regulation scale
Number of participants who score above 80 on an emotion regulation scale | 3-month follow-up
  Number of participants who score above 80 on an emotion regulation scale
Number of participants who score 54 or more on a measure of emotion regulation skills use | 30 days
  The Emotion Regulation Skills Questionnaire is a 27-item measure of the extent to which an individual was able to successfully use emotion regulation skills typically taught in emotion regulation skills training interventions. Scores range from 0 to 108, and higher scores indicate more successful use of emotional regulation skills.
Number of participants who score 54 or more on a measure of emotion regulation skills use | 3-month follow-up
  The Emotion Regulation Skills Questionnaire is a 27-item measure of the extent to which an individual was able to successfully use emotion regulation skills typically taught in emotion regulation skills training interventions. Scores range from 0 to 108, and higher scores indicate more successful use of emotional regulation skills.
Number of participants who score above the clinical range (T score of 70+) on the global severity index of the Symptom Checklist-90 | 30 days
  The Symptom Checklist-90 is A self-report 90-item measure of psychological distress with a T-score range of 30 to 120. Higher scores indicate higher distress.
Number of participants who score above the clinical range (T score of 70+) on the global severity index of the Symptom Checklist-90 | 3-month follow-up
  The Symptom Checklist-90 is A self-report 90-item measure of psychological distress with a T-score range of 30 to 120. Higher scores indicate higher distress.
Number of participants who score 40 or less on a measure of perceived efficacy to abstain from alcohol | 30 days
  Participants will complete the 20-item Alcohol Abstinence Self-Efficacy scale indicating how confident they are in ability to abstain from alcohol in certain situations. Scores range from 20 to 100, with higher scores indicating higher confidence to abstain from alcohol use.
Number of participants who score 40 or less on a measure of perceived efficacy to abstain from alcohol | 3-month follow-up
  Participants will complete the 20-item Alcohol Abstinence Self-Efficacy scale indicating how confident they are in ability to abstain from alcohol in certain situations. Scores range from 20 to 100, with higher scores indicating higher confidence to abstain from alcohol use.
18. Number of participants who score 40 or less on a measure of perceived efficacy to abstain from alcohol | 30 days
  Participants will complete the 20-item Alcohol Abstinence Self-Efficacy scale indicating how confident they are in ability to abstain from alcohol in certain situations. Scores range from 20 to 100, with higher scores indicating higher confidence to abstain from alcohol use
18. Number of participants who score 40 or less on a measure of perceived efficacy to abstain from alcohol | 3-month follow-up
  Participants will complete the 20-item Alcohol Abstinence Self-Efficacy scale indicating how confident they are in ability to abstain from alcohol in certain situations. Scores range from 20 to 100, with higher scores indicating higher confidence to abstain from alcohol use

IPD SHARING:
Plan to Share IPD: No